CLINICAL TRIAL: NCT02031510
Title: Dexmedetomidine as an Adjuvant to Bupivacaine in Transversus Abdominis Plane Block for Laparoscopic Cholecystectomy: Multicentre Study
Brief Title: Dexmedetomidine in Transversus Abdominis Plane Block for Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Anesth-Nov13(2)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Elective Laparoscopic Cholecystectomy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- bupivacaine-dexmedetomidine (Active Comparator): transversus abdominis plane block with bupivacaine 0.25% with dexmedetomidine 1 µg Kg-1
  Interventions: Drug: bupivacaine-dexmedetomidine
- bupivacaine (Active Comparator): transversus abdominis plane block with bupivacaine 0.25%
  Interventions: Drug: bupivacaine
- placebo (Placebo Comparator): Transversus abdominis block with saline 0.9%
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — transversus abdominis plane block with saline 0.9%
  Arms: placebo
Drug: bupivacaine — transversus abdominis plane block bupivacaine 0.25%
  Arms: bupivacaine
Drug: bupivacaine-dexmedetomidine — transversus abdominis plane block with bupivacaine 0.25% with dexmedetomidine 1 µg Kg-1
  Arms: bupivacaine-dexmedetomidine

SUMMARY:
The use of dexmedetomidine as an adjunct to bupivacaine in transversus abdominis plane block will reduce the cumulative morphine consumption after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy, which is a common surgical procedure, is associated with less postoperative pain in comparison to open cholecystectomy. However, this pain needs to be treated adequately to allow early mobilization.

Ultrasound guided transversus abdominis plane (TAP) block is an established technique to manage post laparoscopic cholecystectomy pain. 1 In addition, the use of TAP blocks reduced the need for intraoperative and postoperative opioids and the side-effects associated with their use.

The aim of a TAP block is to deposit local anaesthetic in the plane between the internal oblique and transversus abdominis muscles targeting the spinal nerves in this plane. The innervation to abdominal skin, muscles and parietal peritoneum will be interrupted.

Dexmedetomidine which is an Alpha 2-adrenergic agonist produces analgesia via a non-opioid mechanism and is also known to enhance central and peripheral neural blockades.2 Dexmedetomidine added to bupivacaine or levobupivacaine for brachial plexus block shortens sensory and motor block onset time, extends motor and sensory block durations, and also extends the postoperative analgesia.3, 4

We postulate that the use of dexmedetomidine as an adjunct to bupivacaine in transversus abdominis plane block will reduce the morphine consumption after laparoscopic cholecystectomy.

Based upon previous published data,4 a priori power analysis indicated that 60 patients in each group would be sufficient to detect a 30% reduction in the 24-hours cumulative morphine consumption, which is considered to be of clinical validity, with a type-I error of 0.0167 (0.05/4) and a power of 80%. We added 10% extra patients to compensate for possible dropouts.

All patients will be familiarized with a 10-cm visual analogue scale (VAS) (0= no pain; 10= worst imaginable) to assess the intensity of pain and on the use of the patient-controlled analgesia (PCA).

Monitoring includes non-invasive blood pressure, and electrocardiography, pulse oximetry.

An intravenous infusion of 10 ml kg-1 of Lactated Ringer's solution will be initiated before surgery and will be followed by 5 ml kg-1 hr-1 throughout the procedure.

Anaesthesia technique will be standardized. Anesthesia will be induced by fentanyl of 2-3 µg kg-1, propofol 1.5-2.5 mg kg-1, and rocuronium 0.6 mg kg-1. Tracheal intubation will be carried out at the development of maximum block as monitored by the train-of-four (TOF).

Anesthesia, consisting of a 0.7-1.5 minimum alveolar concentration (MAC) of sevoflurane, will be administered to maintain heart rate (HR) and mean arterial blood pressure (MAP) values below 20% of baseline values. Fentanyl 0.5μg/kg increments will be administered when the HR and MAP values are > 20% of baseline values, despite a target sevoflurane of MAC ≥ 1.5. When the HR and MAP values < 20% of baseline values, the sevoflurane MAC is decreased gradually to 0.7 MAC.

Patients' lungs will be ventilated to achieve a PaCO2 of 35-45 mm Hg. All patients will receive intravenous granisetron 1 mg and lornoxicam 16 mg after the induction of anaesthesia. Rocuronium increments will be given to maintain suppression of the second twitch in the TOF.

The anaesthesiologists who will perform the TAP block and give the anaesthetics will not be involved in the patients' assessment. All other staff in the operating room is unaware of the randomization code.

The TAP block will be performed using ultrasound (SonoSite M-Turbo®, Sonosite, USA) guidance as described by Ra et al

All operations will be performed by the same surgeons. CO2 pneumoperitoneum will be introduced and intra-abdominal insufflation pressure will be limited to 12 mm Hg. After introducing of the four trocars, the patient will be placed in the reverse Trendelenburg position, using up to 30° of head-up tilt. No supplementary dose of muscle relaxant was administered 30 minutes before the end of the surgery.

After desufflation of CO2 pneumoperitoneum, the patient will be returned to the horizontal position and during skin closure; neuromuscular blockade will be antagonized with 50 µg kg-1 neostigmine and 10 µg kg-1 glycopyrrolate. At the last skin suture, desflurane will be discontinued and tracheal extubation will be performed at the discretion of the involved anesthetist in the patient's management.

A standard postoperative analgesic regimen, consisting of 12-hourly intravenous lornoxicam 8 mg, 6-hourly intravenous paracetamol 1 g and intravenous morphine PCA (incremental dose, 1 mg; lockout time, 6-min; a maximum 4-hourly limit, 30 mg), will be used in all patients. If the patient has persistent postoperative nausea and/or vomiting, metoclopramide 10 mg will be administered intravenously when needed.

Other independent investigators who will be blinded to the study protocol and the patient's randomization code will collect the patient's data.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I and II patients
* general anaesthesia

Exclusion Criteria:

* cardiovascular disease
* respiratory disease
* neurological disease
* renal disease
* hepatic disease
* hormonal disease
* pregnancy
* body mass index > 35 kg/m2)
* smokers
* alcohol abuse
* use of antipsychotics
* communication barriers
* local anesthetics allergy
* chronic use of opioids
* use of nonsteroidal anti-inflammatory drug use during the 24 hours immediately preceding surgery
* coagulation disorders
* infection at the needle insertion
* conversion of laparoscopic to open cholecystectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
postoperative 24-hours cumulative morphine consumption | for 24 hours after surgery
  the retrieved postoperative 24-hours cumulative morphine consumption from the PCA pump report

SECONDARY OUTCOMES:
cumulative use of fentanyl | for 2 hours during surgery
  the cumulative doses of fentanyl (from induction through the end of the surgery)
postoperative pain at rest | for 24 hours after surgery
  the degree of postoperative pain at rest at 0.5, 2, 4, 6, 8, 12, 16, 20 and 24 h postoperatively
postoperative pain on movement | for 24 hours aftersurgery
  the degree of postoperative pain at rest at 0.5, 2, 4, 6, 8, 12, 16, 20 and 24 h postoperatively
sedation scores | For 24 hours after surgery
  the degree of sedation scores at 0.5, 2, 4, 6, 8, 12, 16, 20 and 24 h postoperatively
Time to bowel recovery | for 24 hours after surgery
  the times to first flatus, defecation, intake of clear liquid, and solid food tolerated

CONTACTS AND LOCATIONS:
Overall Officials: Abdulmohsen A Al Ghamdi, MD, Principal Investigator — Chairman of Anesthesiology Dept
Locations (2):
- Saudi Arabia (2):
  - King Fahd Hospital of Dammam University, Khobar, Eastern Province
  - Dammam University, Khobar, Eastern Province